CLINICAL TRIAL: NCT05105425
Title: The Effects of Daily Supplementation of Nutriose® on the Fecal Microbiota in Volunteers Over 4 Weeks: a Randomized, Double-blinded, Placebo Conrolled Pilot Study.
Brief Title: The Effects of Daily Supplementation of Nutriose® on the Fecal Microbiota in Volunteers.
Acronym: NUTRIBIOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roquette Freres (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2020-A03403-36
Record Dates: First submitted 2021-07-01; First posted 2021-11-03 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy Male Volunteers
Keywords: Dietary fiber; Microbiota; Stool collection; Shotgun
MeSH Terms: interventions — NUTRIOSE

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A RANDOMIZED, DOUBLE-BLINDED, PLACEBO CONTROLLED PILOT STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUTRIOSE® (Active Comparator): 1 sachet to be taken at breakfast during 4 weeks
  Interventions: Dietary Supplement: NUTRIOSE®
- GLUCIDEX® IT21 (Placebo Comparator): 1 sachet to be taken at breakfast during 4 weeks
  Interventions: Dietary Supplement: GLUCIDEX® IT21 (Placebo)

INTERVENTIONS:
Dietary Supplement: NUTRIOSE® — After randomization (V2 visit), the subjects will consume per os, from V2 to V3, 1 sachet of 15g per day, in the morning, of active formula (NUTRIOSE®) during 4 weeks.
  They will consume 1 sachet in the morning. Powder will have to be mixed with usual beverage of the subject (whatever the type of drink, cold or hot).
  Arms: NUTRIOSE®
Dietary Supplement: GLUCIDEX® IT21 (Placebo) — After randomization (V2 visit), the subjects will consume per os, from V2 to V3, 1 sachet of 15g per day, in the morning, of placebo during 4 weeks.
  They will consume 1 sachet in the morning. Powder will have to be mixed with usual beverage of the subject (whatever the type of drink, cold or hot).
  Arms: GLUCIDEX® IT21

SUMMARY:
The effects of daily supplementation of the NUTRIOSE® on the fecal microbiota. The hypothesis of the study is that the NUTRIOSE® is able to modulate the intestinal microbiota in a positive way, compare to a placebo, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteer,
* Age between 18 and 60 years (limits included),
* BMI between 18.5 and 25 kg/m² (limits included),
* Having a high or a low usual fiber consumption,
* With a usual normal intestinal transit. According to stool questionnaire completed between V1 and V2, mean of the 7 days of completion, maximum 3 stools / day and 5 stools/weeks minimum and with mean normal consistency (from type 3 to type 5 of the BSFS and with a tolerance of 1 to 3 stools in deviation /week) according to the investigator's opinion,
* Non-smoking or with tobacco consumption < 5 cigarettes / day and agreeing to keep his smoking habits unchanged during the all duration of the study,
* Weight stable within ± 5% in the last three months;
* No significant change in food habits or in physical activity in the 3 months before the study and agreeing to keep these habits unchanged throughout the study;
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme
* Agreeing to be registered on the national file of volunteers in biomedical research file.

Exclusion Criteria:

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other metabolic disorder,
* Suffering from gastrointestinal disorders such as celiac disease, Crohn's disease, functional constipation, irritable bowel syndrome or another gastrointestinal found to be inconsistent with the study according to the investigator,
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, uncontrolled cardiac disease, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or another severe disorders found to be inconsistent with the conduct of the study by the investigator,
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient,
* Lactose intolerant,
* Having undergone recent surgical procedure in the past 6 months or planned in the 2 months to come,
* Under treatment which could significantly affect parameter(s) followed during the study according to the investigator or stopped less than 4 weeks before the V1 visit, i.e. medication with impact on intestinal transit such as anti-diarrheal, anti-spasmodic, antidepressants antibiotics, antacids, laxative, antifungal, NSAI, antivomiting, corticoids, opioids, narcotic analgesic and biliary acids chelator, and chronic hormonal treatment started less than 3 months ago (i.e. new method of hormonal contraception, thyroidal trouble treatment)
* Regular intake of dietary supplements or "health foods", or products known to impact intestinal microbiota, containing or rich in prebiotic, probiotic, synbiotics, fiber, fermented milk or yogurt, kefir, ultra-yeast, vitamins and minerals or stopped less than 3 months before the inclusion visit (V1);
* With a current or planned in the next 3 months specific diet (hyper or hypocaloric, vegan, vegetarian…) or stopped less than 3 months before the study,
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded),
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Comparison at V3 of relative abundance of Parabacteroides genus in intestinal microbiota | 4 weeks
  Assessed via Shotgun metagenomics analysis

SECONDARY OUTCOMES:
Comparison at V4 of relative abundance of Parabacteroides genus in intestinal microbiota. | 7 or 8 weeks
  Assessed via Shotgun metagenomics analysis
Comparisons at V3 and V4 of relative abundance of intestinal microbiota (Bacterial species of Parabacteroides genus, Bacteroides genus, Firmicutes phylum, the functional levels of the intestinal microbiota, ...) | 2 weeks
  Assessed via Shotgun metagenomics analysis
Comparisons at V3 and V4 of intestinal parameters : Fecal pH | 2 weeks
  Assessed via laboratory analyse (no unit)
Comparisons at V3 and V4 of intestinal parameters: Fecal short chain fatty acids (SCFA) | 2 weeks
  Assessed via laboratory analyse (µmol/g)
Comparisons at V3 and V4 of intestinal parameters: Secretory immunoglobulin A in feces | 2 weeks
  Assessed via laboratory analyse (mg/g)
The frequency of adverse events | 7 or 8 weeks
  Treatment-Emergent Adverse Events (TEAE), Serious treatment-emergent adverse events (STEAE), TEAEs leading to Investigational Product (IP) discontinuation, Treatment-Emergent Adverse Reaction (TEAR) and gastro-intestinal TEAE.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinical Investigation Unit of Biofortis Paris, Paris
  - Clinical Investigation Unit of Biofortis, Saint-Herblain